CLINICAL TRIAL: NCT03746561
Title: Automatic Diagnosis of Spinal Stenosis on CT With Deep Learning
Brief Title: Automatic Diagnosis of Spinal Stenosis on CT
Acronym: ASSIST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Shanghai East Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Shisheng He, MD, Deputy Director of Orthopedic Department, Shanghai 10th People's Hospital
Other Study IDs: SHSY181022
Record Dates: First submitted 2018-11-07; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Deep Learning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- spinal stenosis: Spinal stenosis is a narrowing of the spaces within your spine, which can put pressure on the nerves that travel through the spine. Spinal stenosis occurs most often in the lower back and the neck.
  Interventions: Diagnostic Test: deep learning

INTERVENTIONS:
Diagnostic Test: deep learning — detect and classify spinal stenosis by deep learning

SUMMARY:
MRI is a common tool for radiographic diagnosis of spinal stenosis, but it is expensive and requires long scanning time. CT is also a useful tool to diagnose spinal stenosis, yet interpretation can be time-consuming with high inter-reader variability even among the most specialized radiologists. In this study, the investigators aim to develop a deep-learning algorithm to automatically detect and classify lumbar spinal stenosis.

DETAILED DESCRIPTION:
MRI is a common tool for radiographic diagnosis of spinal stenosis, but it is expensive and requires long scanning time. CT is also a useful tool to diagnose spinal stenosis, yet interpretation can be time-consuming with high inter-reader variability even among the most specialized radiologists. In this study, the investigators aim to develop a deep-learning algorithm to automatically detect and classify lumbar spinal stenosis. It would be a time-saving workflow if the software can assist the radiologists to detect and locate the suspected lesion.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* with radiologists' CT reports on cervical, thoracic and lumbar stenosis

Exclusion Criteria:

* not applicable (only specific levels with extensive infections, fractures, tumor, high-grade spondylolisthesis would be excluded for analysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal stenosis is a narrowing of the spaces within the spine, which can put pressure on the nerves that travel through the spine. Spinal stenosis occurs most often in the back, the neck, and sometimes the thoracic spine.
  Some people with spinal stenosis may not have symptoms. Others may experience pain, tingling, numbness and muscle weakness. Symptoms can worsen over time.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of deep learning | 1 day
  Diagnostic accuracy of deep learning to determine spinal stenosis compared with radiologists' labels based on CT

SECONDARY OUTCOMES:
Diagnostic Performance of deep learning | 1 day
  Sensitivity, specificity, positive predictive value and negative predictive value of deep learning compared with radiologists' labels based on CT

IPD SHARING:
Plan to Share IPD: Undecided